CLINICAL TRIAL: NCT02947555
Title: Cardiovascular Risk Assesment in Diabetic Patients Via Lens Autofluorecscence Detection
Acronym: CRADILA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Gergő Molnár (Other)
Collaborators: Bajcsy-Zsilinszky Kórház (Unknown); Petz Aladar County Teaching Hospital (Other); Vanderlich Egészségcentrum (Unknown); Semmelweis University Heart and Vascular Center (Other); Polytech Hungaria Kft. (Unknown)
Responsible Party: Sponsor-Investigator, Dr. Gergő Molnár, senior lecturer, University of Pécs, University of Pecs
Organization: University of Pecs (Other)
Other Study IDs: PTEBEL 01/2015
Record Dates: First submitted 2016-09-22; First posted 2016-10-28 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Diabetic Patients With/Without Atherosclerotic Diseases
Keywords: diabetes mellitus; atherosclerosis; AGE; lens autofluorescence
MeSH Terms: conditions — Diabetes Mellitus; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- DM+/AT+: Patients with type 2 diabetes mellitus and atherosclerotic event in history
  Interventions: Other: Non interventional
- DM+/AT-: Patients with type 2 diabetes mellitus without atherosclerotic event in history
  Interventions: Other: Non interventional
- DM-/AT+: Non-diabetic patients with atherosclerotic event in history
  Interventions: Other: Non interventional
- DM-/AT-: Non-diabetic patients without atherosclerotic event in history
  Interventions: Other: Non interventional

INTERVENTIONS:
Other: Non interventional

SUMMARY:
The rate of lens autofluorescence will be compared in diabetic and non diabetic patients with/without atherosclerotic vascular diseases to evaluate if it is associated with the risk of cardiovascular diseases.

DETAILED DESCRIPTION:
The rate of lens autofluorescensce is associated with the accumulation of advanced glication endproducts (AGE).The concetration of AGE increases with age but is also higher in diabetic patients. There is evidence that diabetes could be diagnosed via the detection of lens autofluorescence. The investigators are planning a cross sectional clinical trial to evaluate if the rate of lens autofluorescence could be associated with the clinical appearance of atherosclerotic vascular diseases in diabetic/non-diabetic patients and in patients who already had atherosclerotic vascular events and patients without previous atherosclerotic events. The cardiovascular and metabolic histoty of patients will be evaluated using a questionaire. Antropometrical data, blood pressure, heart rate, glucose metabolism, serum lipid profile, CRP, serum creatinine (eGFR) will be assased. ClearPath DS-120 biomicroscopical optical system (Freedom Meditech, San Diego, CA, USA) will be used for the measurment of lens autofluorescence. The measurement will be performed on one eye. Data of the different patient groups will be compared using ANOVA, a value of p<0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years either wit type 2 diabetes or non-diabetic, either having atherosclerotic vascular events in history or not (ACS, angina pectoris, stroke, TIA, clinically symptomatic PAD, atherosclerosis based amputation, stent implantation, angiplasty) Diabetes present for more than 1 year.

Exclusion Criteria:

* patient did not signe informed consent
* cataract
* after cataract operation, after optical operation, after sclera injury
* fluorescein angiograpy performed in 6 months
* diseases affecting the eye surface( sleritis, Sjogren sy)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-75 years either wit type 2 diabetes or non-diabetic, either having atherosclerotic vascular events in history or not (ACS, angina pectoris, stroke, TIA, clinically symptomatic PAD, atherosclerosis based amputation, stent implantation, angiplasty) Diabetes present for more than 1 year.
Sampling Method: Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2016-05-01; Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Association of lens autofluorescence with atherosclerotic vascular events | 2 years
  Measurement of the autofluorescence of lens proteins and assessement of its association with the occurrance of atherosclerotic vascular events

SECONDARY OUTCOMES:
Association of lens autofluorescence with the perscene of diabetes | 2 years
  Measurement of the autofluorescence of lens proteins and assessement of its association with the persence of diabetes type 2 diabetes
Association of lens autofluorescence with renal function | 2 years
  Measurement of the autofluorescence of lens proteins and assessement of its association with renal function (eGFR)
Association of lens autofluorescence with glucose metabolism parameteres | 2 years
  Measurement of the autofluorescence of lens proteins and assessement of its association with glucose metabolism parameteres (ex. HBA1C, HOMA IR)
Association of lens autofluorescence with lipid profile | 2 years
  Measurement of the autofluorescence of lens proteins and assessement of its association with serum lipid values (serum total cholesterol, triglycerids, LDL, HDL)
Association of lens autofluorescence with CRP | 2 years
  Measurement of the autofluorescence of lens proteins and assessement of its association with CRP level
Association of lens autofluorescence with antropoetric parameters | 2 years
  Measurement of the autofluorescence of lens proteins and assessement of its association with antropometric parameteres (body weight, height, BMI, waist-hip ratio)

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of Medicine and Nephrological Center, Pécs, Baranya, Hungary